CLINICAL TRIAL: NCT01795469
Title: Abdominal and Lower Extremity Compression During Tilt Table Testing in Adolescent POTS Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Geoffrey Heyer, Assistant Professor, Nationwide Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB13-00033 (NCH IRB number)
Record Dates: First submitted 2013-02-18; First posted 2013-02-20 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Postural Orthostatic Tachycardia Syndrome (POTS); Syncope
Keywords: POTS; Orthostatic; Adolescent
MeSH Terms: conditions — Postural Orthostatic Tachycardia Syndrome; Syncope

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Abdominal and LE compression (Experimental): Zoex compression garment during tilt testing (all straps)
  Interventions: Device: Zoex compression garment
- abdominal compression only (Experimental): Zoex compression garment use during tilt table testing (straps 4 and 5 fastened around thighs and abdomen)
  Interventions: Device: Zoex compression garment
- Lower extremity compression only (Experimental): Zoex compression garment use during tilt table testing (straps 1-4, lower extremity and thighs, fastened)
  Interventions: Device: Zoex compression garment

INTERVENTIONS:
Device: Zoex compression garment — 5-strap compression of abdomen, thighs and legs

SUMMARY:
Postural orthostatic tachycardia syndrome (POTS) is a common cause of orthostatic intolerance in adolescents and adults. Compression stockings are commonly recommended as a treatment modality for POTS, but the effects of abdominal and lower extremity compression during tilt table testing have not been measured in adolescent patients. The aims of our study are to compare heart-rate changes and symptom onset during tilt table testing (a) with and without abdomen/lower extremity compression and (b) with abdominal compression only versus lower extremity compression only. During phase 1, 20 adolescents with POTS will undergo up to 10 minutes of tilt without compression (trial #1), a repeat study of up to 10 minutes with full compression (trial #2), and a third study without compression up to 10 minutes (trial #3). Compression will be performed using the non-inflatable Zoex anti-shock garment. During study phase 2, an additional 20 adolescent POTS patients will undergo up to 10 minutes of tilt without compression (trial #1), a repeat study of up to 10 minutes with abdominal compression only [n=10] or lower extremity compression only [n=10] (trial #2), and a third study repeated without compression up to 10 minutes (trial #3). To limit compression to the abdomen only, we will use the Zoex garment strap numbers 4 and 5 (thigh and abdomen) without straps 1-3 (lower extremities). For lower extremity-only compression, we will use Zoex garment straps 1-4 (lower extremity and thigh) without strap 5. Data collected will include mean and peak heart rates and timing of symptoms with each trial. A paired-samples t-test will be used to compare mean heart rates between trials for each study phase. Hazard analyses will be used to assess time-based endpoints.

ELIGIBILITY:
Inclusion Criteria:

1. Age 12-19 years
2. POTS diagnosis
3. English speaking -

Exclusion Criteria:

1. Somatic, cognitive, or psychiatric disorder that could prevent safe tilt table testing
2. Medications that cannot be stopped/held safely for the procedure, but can cause or exacerbate orthostatic intolerance -

Ages: 12 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2013-02; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Heart-rate elevation | Comparison between tilt table trials of up to 10 minutes duration without and with abdominal and/or lower extremity compression

SECONDARY OUTCOMES:
Symptom onset | Comparison between tilt table trials of up to 10 minutes duration witout and with abdominal and/or lower extremity compression

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, neurology outpatient clinic, Columbus, Ohio, United States

REFERENCES:
- [Result] Heyer GL. Abdominal and lower-extremity compression decreases symptoms of postural tachycardia syndrome in youth during tilt table testing. J Pediatr. 2014 Aug;165(2):395-7. doi: 10.1016/j.jpeds.2014.04.014. Epub 2014 May 17. PMID 24840763